CLINICAL TRIAL: NCT01981785
Title: Investigation of Molecular, Genetic and Cellular Mechanisms of Human Immune Disorders and Deficiencies
Brief Title: Investigation of Immune Disorders and Deficiencies
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: O & O Alpan LLC (Other)
Responsible Party: Principal Investigator, Oral Alpan, Principal Investigator, O & O Alpan LLC
Other Study IDs: 12-CFCT-04
Record Dates: First submitted 2013-05-06; First posted 2013-11-13 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Primary Immune Deficiencies; Autoimmune Diseases; Inflammatory Diseases; Common Variable Immune Deficiencies; Hypogammaglobulinemia
Keywords: Primary immune deficiencies; Autoimmune diseases; Inflammatory diseases; Common variable immune deficiencies; Primary Immunodeficiencies; Immunoglobulin; IgG; IVIG; Recurrent Infections
MeSH Terms: conditions — Primary Immunodeficiency Diseases; Autoimmune Diseases; Agammaglobulinemia; Reinfection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Immune deficiencies/Immune disorders: Patients with abnormal immune responses or potential primary immune deficiencies or immune disorders (allergies, autoimmune diseases) will be enrolled as the study group.
- No prior immune abnormalities: Patients with no prior immune abnormalities will be enrolled as the control group.

SUMMARY:
The immune system is an intricate system comprised of specialized cells, proteins, tissues and organs. Proper functioning is critical to the body's ability to defend itself against harmful pathogens. Immunological disorders and deficiencies are defects in the immune system that lead to abnormal immune responses. Abnormal immune responses could be derived from immune deficiencies, dysregulations or hypersensitivities.

The overall goal of this research study is to identify the mechanisms of primary immune deficiencies and immune disorders at the genetic, cellular and molecular level, using novel analytic techniques to be performed on immune cells derived from blood samples. The knowledge gained from the aims of this study could lead to better diagnostics and identify novel targets for therapeutic interventions.

DETAILED DESCRIPTION:
Primary immunodeficiency diseases (PID) represent a class of disorders in which there is an instrinsic defect in the human immune system. The PID could be caused by defects or perturbations in either the innate or adaptive immune cells, such as B cell defects which result in lack of antibodies. Research in this topic remains a difficult feat due factors such as genetic heterogeneity and the gene-environment interface. Limitations of standard of care testing leads to many patients with immunological problems to be undiagnosed. In addition to the variety of primary immune deficiencies, there are large number of immune system disorders due to various perturbations in the immunological components that cause diseases with much greater prevalence such as autoimmune diseases, lymphoproliferative diseases, chronic inflammation and certain cancers. The causes of these immune disorders are typically more complex than PID but there are also many overlaps in immune hyper-activation and deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Subject is greater than or equal to 1 day of age and less than or equal to 100years of age
* Signed Informed Consent/Assent
* Subject is able and willing to comply with study protocol requirements
* From clinical or blood laboratory findings subject has evidence of immune abnormalities (or no immune abnormalities in the case of controls) or immune-mediated disease.

Exclusion Criteria:

* Risk factors for donating blood (such as anemia or blood clotting disorders)

Min Age: 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with abnormal immune responses or potential PID or immune disorders (allergies, autoimmune diseases) will be enrolled as the study group and patients with no prior immune abnormalities will be enrolled as the control group.
Sampling Method: Non-Probability Sample
Enrollment: 343 (Actual)
Dates: Start 2012-12; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Genetic variants | 10 years
  To elucidate genetic variants associated with various previously identified immune disorders to include but not limited to immune dysregulations, hypersensitivities, inflammatory conditions and deficiencies.

SECONDARY OUTCOMES:
Pathogenesis | 10 years
  To further elucidate pathogenesis of previously discovered immune disorders or subjects with suspected allergic/immunological disorders using cell surface and intracellular staining techniques using flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Oral Alpan, MD, Principal Investigator — O & O Alpan LLC
Locations (1):
- O&O Alpan LLC, Fairfax, Virginia, United States

REFERENCES:
- See also: Related Info — http://oandoalpan.com/